CLINICAL TRIAL: NCT03640390
Title: Dexmedetomidine Versus Magnesium Sulfate Infusion During Spinal Anesthesia for Lower Abdominal Surgery
Brief Title: Dexmedetomidine Versus Magnesium Sulfate Infusion During Spinal Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-112-2017
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group (Experimental): This group will receive dexmedetomidine infusion at a rate of 0.5 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine
- Magnesium Sulphate group (Active Comparator): This group will receive Magnesium Sulphate infusion at a rate of 15 mg/Kg/hour
  Interventions: Drug: Magnesium Sulphate
- Saline group (Placebo Comparator): This group will receive normal saline infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — This group will receive Dexmedetomidine infusion at a rate of 0.5 mcg/kg/hour.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Magnesium Sulphate — This group will receive Magnesium sulphate infusion at a rate of 15 mg/Kg/hour
  Arms: Magnesium Sulphate group
Drug: Normal saline — This group will receive normal saline infusion
  Arms: Saline group

SUMMARY:
The aim of this work is to compare the hemodynamic and analgesic properties of Dexmedetomidine and Magnesium sulphate infusion in lower abdominal surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a relatively new alpha 2 adrenergic receptor agonist with a higher α2/α1 selectivity ratio of 1620:1 that provides analgesic and anesthetic effects . Dexmedetomidine has various clinical uses in anesthesia such as sedation, and prolongation of the duration of postoperative analgesia when used as an adjuvant through intrathecal, epidural, or intravenous routes.

Magnesium sulphate is another commonly used drug in anesthesia. Magnesium sulphate suppresses nociceptive impulses through inhibition of voltage-gated calcium channels and through antagonism of the N-methyl D-aspartate (NMDA) receptors.

Although both drugs were reported to prolong the duration of spinal anesthesia, no studies to the best of our knowledge had compared the analgesic and hemodynamic profile of both drugs when used as intravenously during spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 65 years.
* Scheduled for lower abdominal surgery.

Exclusion Criteria:

* Systolic blood pressure less than 100 mmHg
* Coagulation disorders
* History of heart failure
* Mitral or Aortic stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  Duration of analgesia after the operation defined as the time till the first analgesic request by the patient

SECONDARY OUTCOMES:
Systolic blood pressure | 6 hours
  Systolic blood pressure measured in mmHg
Diastolic blood pressure | 6 hours
  Diastolic blood pressure measured in mmHg
Heart rate | 6 hours
  The number of heart beats per minute
Onset of sensory block | 30 minutes after spinal anesthesia
  The time needed to have complete sensory block after spinal anesthesia measured in minutes
Onset of motor block | 30 minutes after spinal anesthesia
  The time needed to have complete motor block after spinal anesthesia measured in minutes
Duration of motor block | 12 hours
  The time needed for recovery of motor motor after spinal anesthesia measured in hours
Ramsay Sedation Scale | 12 hours after spinal anesthesia
  A scale used for assessment of sedation level ranges from 1 (combative) to 6 (unarousable)

CONTACTS AND LOCATIONS:
Overall Officials: Inas Farouk, Lecturer, Study Director — Lecturer of anesthesia
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No